CLINICAL TRIAL: NCT01840345
Title: The Role of N-acetyl-l-cysteine (NAC) as an Adjuvant to Opioid Treatment in Patients With Chronic Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM14748
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Neuropathic Pain
Keywords: uncontrolled; neuropathic pain
MeSH Terms: conditions — Neuralgia | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- N-acetyl-L-cysteine (Experimental): n-acetyl-l-cysteine 1200 mg BID x 4 weeks
  Interventions: Drug: N-acetyl-l-cysteine

INTERVENTIONS:
Drug: N-acetyl-l-cysteine — 1200 mg BID x 4 weeks
  Other Names: NAC

SUMMARY:
This study will test whether treatment with N-acetyl-L-cysteine (NAC) is safe and decreases pain in patients with chronic neuropathic pain. The investigators hypothesize that NAC will be a useful adjunct to opioid treatment in chronic neuropathic pain.

DETAILED DESCRIPTION:
This is an open-label study to evaluate the safety and efficacy of N-acetyl-L-cysteine in patients with Chronic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* non-cancer neuropathic pain
* stable dose of opioids for pain
* using breakthrough pain meds
* still with persistent pain per VAS

Exclusion Criteria:

* pregnant or nursing
* serious medical or psychiatric illness (including uncontrolled hypertension)
* active stomach ulcer, history or seizures or asthma
* breakthrough pain meds other than opioids
* using illicit drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-01; Primary Completion 2017-03-01 (Actual); Study Completion 2017-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dace S Svikis, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-acetyl-L-cysteine
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: One patient did not complete study so was not included in efficacy analysis
Arm/Group | N-acetyl-L-cysteine
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use
Description: The amount of opioid medication used was recorded. Then, it was converted to morphine equivalents (https://www.cms.gov/Medicare/Prescription-Drug-Coverage/PrescriptionDrugCovContra/Downloads/Opioid-Morphine-EQ-Conversion-Factors-March-2015.pdf). Opioid use was measured over a 2-week baseline period. Then, the average opioid medication use/week was calculated. This was compared to the average opioid medication use/week after 4 weeks of NAC.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: morphine equivalent dose
Arm/Group | N-acetyl-L-cysteine
Number analyzed (Participants) | 10
morphine equivalent dose
  Baseline | 101.24 (89.93)
  4 weeks | 104.56 (96.66)

2. Secondary Outcome: Pain
Description: Pain intensity will be measured by using the 100-point Visual Analogue Scale, a 100-mm horizontal line with anchors of "no pain at all" (at 0) and "worst pain imaginable" (at 100mm) on which patients' pain intensities are measured.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: mm on 100 mm scale
Arm/Group | N-acetyl-L-cysteine
Number analyzed (Participants) | 10
mm on 100 mm scale
  Baseline | 6.38 (1.58)
  4 weeks | 5.95 (1.96)

3. Secondary Outcome: Mood
Description: Mood will be assessed by using the Patient Health Questionnaire (PHQ-9), a validated 9-question assessment of depression with total scores ranging from 0-27. Higher score = worse depression.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetyl-L-cysteine
Number analyzed (Participants) | 10
units on a scale
  Baseline | 10.4 (4.9)
  4 weeks | 9.7 (6.5)

4. Secondary Outcome: Stress
Description: Stress will be measured by the Perceived Stress Scale ((PSS), a 10-item instrument for measuring the perception of stress, with total scores ranging from 0-40. Higher scores = higher perceived stress
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetyl-L-cysteine
Number analyzed (Participants) | 10
units on a scale
  Baseline | 21.5 (3.6)
  4 weeks | 16.6 (1.4)

ADVERSE EVENTS:
Time Frame: A physical examination was done at Baseline. Then, adverse events were assessed at each study visit throughout the study and follow-up periods.
Description: All participants were asked about side effects and adverse events on a weekly basis, and any adverse events reported by the patients were evaluated by study staff.
Arm/Group | N-acetyl-L-cysteine
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 10/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetyl-L-cysteine (N=11)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Gastroesophageal reflux (Gastrointestinal disorders) | 5 (6)
Loss of appetite (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Itching (Skin and subcutaneous tissue disorders) | 2 (2)
Sweating (Endocrine disorders) | 2 (2)
Sleepy (Nervous system disorders) | 1 (2)
chronic colonic ileus (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
All adverse events reported regardless of causality

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT01840345/Prot_SAP_000.pdf